CLINICAL TRIAL: NCT03141905
Title: Can a Sick-Day Protocol to Improve Outcomes in Chronic Kidney Disease?
Brief Title: Sick-Day Protocol to Improve Outcomes in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jeffrey Fink, Division Head, General Internal Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HP-00069775
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Safety Issues; Chronic Kidney Diseases
Keywords: patient safety; self-management; remote monitoring
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sick-Day Protocol (Active Comparator): Sick-Day Protocol (instructions for holding and resumption of certain medicines in the event of dehydrating illness) and IVRSDRS weekly remote monitoring
  Interventions: Other: Sick-Day Protocol
- Usual Care (Placebo Comparator): Standard clinical care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Sick-Day Protocol — Sick-Day Protocol (instructions for holding and resumption of certain medicines in the event of dehydrating illness) and IVSDRS weekly remote monitoring
  Arms: Sick-Day Protocol
Other: Usual Care — Standard clinical care
  Arms: Usual Care

SUMMARY:
The benefits of renin angiotensin system (RAS) blockers and diuretics for blood pressure control are well-established in chronic kidney diseases (CKD) patients; however, these agents may become hazardous on "sick-days" that lead to volume depletion (dehydration), and increase the risk of kidney function loss and acute kidney injury (AKI). It is not known how frequent significant sick-days occur in CKD patients, or whether a patient self-managed Sick-Day Protocol (SDP) that temporarily holds RAS blocker, diuretics, or other high risk medication in an effort to preserve renal function, or prevent AKI. The purpose of the study is to asses if a SDP, monitored remotely with a weekly automated phone survey , can improve outcomes in CKD (such as slow renal function loss and AKI episodes) and reduce preventable service utilization versus usual care.

DETAILED DESCRIPTION:
Hypothesis: implementing a self managed "Sick-Day Protocol" with telephone monitoring via interactive voice survey dial-response system (IVSDRS) in CKD patients taking RAS blockers, diuretics, metformin, or NSAIDs, will safely slow renal function loss, reduce the incidence of acute kidney injury, and prevent urgent health utilization; in comparison to usual care.

Study Design: 6-month randomized trial of Sick-Day Protocol vs usual care

Randomization: In-block randomization stratified by use (with or without any other qualifying medication) vs non-use of RAS blocker (with any other qualifying medication)

Intervention: Sick-Day Protocol (instructions for holding and resumption of certain medicines in the event of dehydrating illness), IVRSDRS remote monitoring, augmented laboratory monitoring, and decision support from the VA Renal Inter-disciplinary Safety clinic (RISC)

Study Population: Veterans across the VA Maryland Health Care System (VAMCHS) with a current prescription for any type of RAS blocker, Diuretic, Metformin or NSAID.

Study Site: Baltimore VA Medical Center (BVAMC), VA Geriatrics Research Education and Clinical Center (GRECC).

Specific Aims 1: Conduct a pragmatic trial comparing the renal function decline, incidence of AKI, and urgent service utilization in eligible CKD patients provided with a self-managed Sick-Day Protocol versus comparable patients receiving usual care.Specific Aim 2: Determine the incidence of sick-days in the intervention arm using remote IVSDRS monitoring and end-of-study survey of all participants. Specific Aim 3: Evaluate intervention arm participants' usage of, and adherence to, the Sick-Day Protocol with remote IVSDRS monitoring.

Study Measurements: laboratory-measured renal function, and patient- reported safety events obtained per IVSDRS protocol. Emergency department (ED) visits, hospitalization, renal progression, incidence of ESRD, and death will be measured in both groups along with patient satisfaction.

Primary outcomes: 6-month change in renal function (eGFR), incidence of AKI episodes (including ICD-10 code designated, and detectable creatinine-based changes in renal function usingRIFLE criteria), preventable/urgent service utilization (to be ascertained using VA EHR review)

Secondary outcomes: Determination of incidence of sick-day events (IVSDRS reporting, and end-of-study self-report).

Tertiary:Adherence to self-management Sick-Day Protocol (based on IVSDRS reporting)

Analytic plans: Comparison between intervention and usual care participants of 6-month renal function change, and frequency of AKI and hospitalization using generalized linear models and Poisson regression methods, respectively. Similar regression methods will be used to determine the adjusted frequency rate of sick-day incidents and participant response to sick-days.

Public Health Relevance: Introduction of a self-management Sick-Day Protocol in conjunction with coordinated care and IVSDRS surveillance can be an innovative strategy to improve renal outcomes and reduce preventable service utilization.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with prescription for any type of RAS blocker, diuretic, Metformin or NSAID

Exclusion Criteria:

* Expected death or dialysis within 6 months
* No home or cellular telephone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Fink JC, Maguire RM, Blakeman T, Tomlinson LA, Tomson C, Wagner LA, Zhan M. Medication Holds in CKD During Acute Volume-Depleting Illnesses: A Randomized Controlled Trial of a "Sick-Day" Protocol. Kidney Med. 2022 Jul 31;4(9):100527. doi: 10.1016/j.xkme.2022.100527. eCollection 2022 Sep. PMID 36046613

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sick-Day Protocol | Usual Care
Started | 176 | 166
Completed | 152 | 147
Not Completed | 24 | 19
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 3 | 7
Not completed — Randomized, but did not receive intervention. Withdrew prior to baseline visit. | 17 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sick-Day Protocol | Usual Care | Total
Number analyzed (Participants) | 159 | 156 | 315
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 37 | 66
  >=65 years | 130 | 119 | 249
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 152 | 149 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 158 | 155 | 313
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 100 | 99 | 199
  White | 58 | 56 | 114
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 159 | 156 | 315
eGFR [Mean (Standard Deviation); unit: ml/min/1.73m^2] — Population: Baseline creatinine/eGFR missing for 4 study participants, 3 in the usual care arm, and 1 in the intervention arm.
  ml/min/1.73m^2
    number analyzed (Participants) | 158 | 153 | 311
    (all) | 43.110 (13.128) | 43.783 (13.018) | 43.441 (13.057)

OUTCOME MEASURES:

1. Primary Outcome: Change in Renal Function From Baseline to Study Completion;
Description: Laboratory measurement of creatinine at study entry and completion
Time Frame: 6 months (enrollment to study completion)
Population: 280 participants with complete laboratory data collection
Measure: Median (95% Confidence Interval); unit: mg/dL
Arm/Group | Sick-Day Protocol | Usual Care
Number analyzed (Participants) | 140 | 140
mg/dL | 0.01 [-0.11 to 0.22] | 0.02 [-.010 to 0.21]

2. Secondary Outcome: Acute Kidney Injury Incidents
Description: Participants with abrupt changes in renal function as determined by EHR post-study review of new AKI ICD-10 codes, and for-cause lab ambulatory lab testing using RIFLE criteria
Time Frame: 6 months (enrollment to study completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Sick-Day Protocol | Usual Care
Number analyzed (Participants) | 159 | 156
Participants
  AKI ICD-10 code on ED visit or admission | 4 | 4
  50% increase in Creatinine | 1 | 0

3. Secondary Outcome: ER Use and Hospitalization
Description: Participants with urgent service utilization including emergency department, hospitalization, and urgent care.
Time Frame: 6 months (enrollment to study completion)
Measure: Count of Participants; unit: Participants
Arm/Group | Sick-Day Protocol | Usual Care
Number analyzed (Participants) | 159 | 156
Participants
  Hospitalization | 29 | 23
  Emergency Room | 35 | 30
  Urgent Care | 5 | 5

4. Other Pre Specified Outcome: Determination of Sick-day Incidents
Description: Participants reporting sick-days via IVSDRS and end-of study visit survey ascertainment.
Time Frame: 6 months from enrollment in study
Population: 299 participants who completed all study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Sick-Day Protocol | Usual Care
Number analyzed (Participants) | 152 | 147
Participants | 29 | 20

5. Other Pre Specified Outcome: Adherence to the Self-management Sick-day Protocol
Description: Frequency of Sick-Day qualifying illnesses reported. (Note: this outcome is N/A for the usual care group)
Time Frame: 6 months (enrollment to study completion)
Population: Sick-Day Protocol group
Measure: Number; unit: count of qualifying illnesses
Arm/Group | Sick-Day Protocol
Number analyzed (Participants) | 159
count of qualifying illnesses
  Followed Sick-Day Protocol instructions | 14
  Did not stop medicines | 12
  Stopped other medicines in addition to SDP qualifying. | 6

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sick-Day Protocol | Usual Care
All-Cause Mortality (participants affected / at risk) | 3/159 | 2/156
Serious Adverse Events (participants affected / at risk) | 0/159 | 0/156
Other Adverse Events (participants affected / at risk) | 7/159 | 3/156
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sick-Day Protocol (N=159) | Usual Care (N=156)
Initiation of Hemodialysis (Renal and urinary disorders) | 1 (1) | 1 (1)
Lab Alert: Glucose ≥ 499 mg/dL (Endocrine disorders) | 1 (1) | 2 (2)
Lab Alert: Potassium ≥ 6.1 mEq/dL (Cardiac disorders) | 3 (3) | 1 (1)
Lab Alert: Hemoglobin ≤ 7.5 g/dL (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lab Alert: Chloride ≥ 115 mEq/dL (Renal and urinary disorders) | 2 (2) | 0 (0)
Lab Alert: Co2 ≤ 15 mEq/L (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic in-person visits were suspended on 3/12/2020 per institution and IRB mandate. Study lab measurements were delayed for 24 participants and not completed for 8 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03141905/Prot_SAP_000.pdf